CLINICAL TRIAL: NCT06262750
Title: Evaluation of Safety and Efficacy of Anticoagulation Treatment in Patients With Splanchnic Vein Thrombosis: SAPIENT Study
Acronym: SAPIENT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DE STEFANO VALERIO, Full Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 00375/23
Record Dates: First submitted 2023-11-07; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Splanchnic Vein Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective single-centre, observational study with medical products. Patients with a medical history of SVT will be observed for at least 24 months after inclusion. The study will begin when the patient is referred to our centre for SVT and will end at the 24-month follow-up or at the occurrence of a study outcome event, or in case of Death OBJECTIVE: To prospectively define the incidence of recurrent thrombosis and bleeding events during anticoagulant therapy in patients with diagnosed SVT, regardless of whether they will be hospitalized or treated as outpatients

ELIGIBILITY:
Inclusion Criteria

* age ≥ 18 years
* ability to provide informed consent;
* confirmed diagnosis of deep vein thrombosis involving splanchnic veins in liver cirrhosis (with or without hepatocarcinoma);
* confirmed diagnosis of deep vein thrombosis involving splanchnic veins in absence of liver cirrhosis (with or without portal cavernoma);
* pregnant patients will be eligible for inclusion in the study;
* ongoing anticoagulant treatment with vitamin K-antagonists (VKA), direct oral anticoagulants (DOAC), low molecular weight heparin (LMWH), fondaparinux

EXCLUSION CRITERIA

* splanchnic vein tumor thrombosis;
* absence of antithrombotic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients referred to the Fondazione Policlinico Universitario Agostino Gemelli IRCCS for SVT, either as inpatients or outpatients, and requiring anticoagulant therapy will be eligible for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidenze of bleedings events | through study completion, an average of 1 year
  Bleeding events will be classified according to ISTH definition, as follows:major bleedings,clinically relevant non-major bleedings (CRNMB), minor bleedings
Incidence of venous and arterial thromboembolic events | through study completion, an average of 1 year
  All venous and arterial thromboembolic (VTE and ATE) events during the study period will be registered and counted
Rate of progress /stable /regressive | every six months, up to 2 years
  To evaluate the impact of anticoagulation therapy on SVT, all enrolled patients will undergo imaging test (doppler ultrasound, contrast-enhanced CT or MR angiography).
incidence of liver related events | through study completion, an average of 1 year
  To evaluate the onset of liver-related events (variceal bleeding, ascites, bacterial infections, and hepatic encephalopathy), all enrolled patients will be clinically assessed

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Servizio e DH Ematologia, Rome, Italy